CLINICAL TRIAL: NCT00349895
Title: Healthy Endothelial Accelerated Lining Inhibits Neointimal Growth. A Clinical, Multi-center, Prospective, Non-Randomized Study
Brief Title: Healthy Endothelial Accelerated Lining Inhibits Neointimal Growth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrbusNeich (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEALING IIb
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis
Keywords: Percutaneous Transluminal Coronary Angioplasty; Stent implantation
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Coronary stent implantation — Percutaneous Coronary Intervention

SUMMARY:
This is a multi-center, prospective, non-randomized study. Approximately 90 patients from up to 16 centers will be entered in the study. Patients will be followed clinically for up to 5 years post-procedure. All patients will have a repeat angiography at 6 months follow-up.

The primary objective of this study is to evaluate the safety and effectiveness of the Genous Bio-engineered R stentTM in conjunction with optimal statin therapy (80mg of atorvastatin), in the treatment of elective patients with up to two de novo native coronary artery lesions. The Genous stent received CE mark for the intended indication in August 2005

DETAILED DESCRIPTION:
Currently available coronary stents are prone to thrombosis and restenosis. It is believed that the accelerated re-establishment of a functional endothelial layer on damaged stented vascular segments may help to prevent potentially serious complications by providing a barrier to circulating cytokines, and by the ability of endothelial cells to produce substances that passivate the underlying smooth muscle cell layer.

By recruiting the patient's own EPCs to the site of vascular injury (e.g. the site of a coronary stent implant), an acceleration of the normal endothelialization process would occur. It is theorized that the rapid establishment of a functioning endothelial layer may promote the transformation of the injured site to a healthy state. For example, in the case of coronary stent implantation, rapid re-endothelialization may reduce inflammation, thrombosis and potentially eliminate restenosis.

The influences of EPC recruitment and reendothelialization on restenosis range from the effects on the vascular repair response, to the prevention of platelet aggregation and activation, angiogenesis, and enhancement of vasomotor response. Recently it has been shown that the integrity and functional activity of the endothelial monolayer play a crucial role in the prevention of atherosclerosis. However, risk factors for coronary artery disease such as age, hypertension, hypercholesterolemia, and diabetes reduce the number and functional activity of these circulating EPCs, thus limiting the regenerative capacity. The impairment of stem cells by risk factors in CAD patients may contribute to the limited regenerative capacity of diseased endothelium, as well as to atherogenesis and atherosclerotic disease progression. Therefore, relating the number and function of circulating EPCs to the functional outcome of stent technology is crucial to identify a beneficial effect on in-stent restenosis formation and vascular (dys) function.

The HEALING FIM and HEALING II clinical studies sought to define the safety and efficacy of a stent designed to sequester circulating endothelial progenitor cells to the luminal surface of the stent struts by an anti-CD34 antibody coating, thereby promoting reendothelialization of the coronary stent and the vascular healing response following stent deployment. Enhanced vascular healing will reinstate vascular integrity, prevent platelet aggregation and sub-acute in-stent thrombosis, reinstate vasoreactivity and inhibit restenosis formation. In the HEALING II study, a correlation was found between EPC levels and angiographic/IVUS outcomes in patients receiving the Genous stent. Patients with normal EPC titers had significantly less in-stent late loss compared to those with low EPCs (0.53 vs 1.02mm). This is consistent with the results from drug eluting stent trials, thereby establishing proof of concept of the EPC capturing technology, provided adequate EPC target cell population is available.

There are several animal studies demonstrating that statin therapy was associated with a 2.5 to 3 fold increase of circulating EPCs leading to accelerated reendothelialization, vascular repair and improved angiogenesis. In addition, Dimmeler and co-workers found similar results in a small cohort of cardiovascular patients receiving atorvastatin therapy (n=7, Circulation 2001), suggesting an angiotrophic effect of atorvastatin therapy in addition to its previously defined pleiotrophic properties. Similarly, Drexler and co-workers described similar EPC recruiting properties of simvastatin in CAD patients unrelated to/ irrespective of LDL reduction (n=10, Circulation 2005).

The current study seeks to confirm the safety and optimize the effectiveness of the EPC capture technology (Genous Bio-engineered R stent) by incorporating a high dose statin therapy, specifically atorvastatin 80mg, for at least two weeks prior to the index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 85 years of age;
2. Symptomatic ischemic heart disease (CCS class 1-4, Braunwald class IB, IC, and/or objective evidence of myocardial ischemia);
3. Treatment of 1 or 2 de novo lesions;
4. Target lesion(s) is(are) located in a native coronary artery, which can be covered by one single stent of maximum 33 mm; The coronary artery lesion should be ≤27 mm in length (a margin of 3mm proximal and 3mm distal is recommended) and should be entirely covered by one single Genous Bio-engineered R stentTM . If predilation of the lesion is visually deemed necessary it should be performed prior to measuring the length of the lesion.
5. Reference vessel diameter ≥ 2.5 and ≤ 3.75 mm by visual estimate;
6. Acceptable candidate for coronary artery bypass surgery (CABG);
7. Target lesion stenosis is ≥50% and <100% (minimum TIMI flow I at the time of the PCI procedure) (visual estimate);
8. The patient is willing to comply with the specified follow-up evaluation;
9. The patient has been informed of the nature of the study agrees to its provisions and has provided written informed consent, approved by the appropriate Ethics Committee (EC).

Exclusion Criteria:

General exclusion criteria:

1. Women who are pregnant or women of childbearing potential who do not use adequate contraception;
2. A Q-wave or non-Q-wave myocardial infarction within 72 hours preceding the index procedure, unless the CK and CK-MB enzymes or Troponin levels are less than twice the Upper Normal Limit;
3. Impaired renal function (creatinine > 3.0 mg/dl or 265 µmol/l);
4. Any patient who has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3 or a WBC of < 3,000 cells/mm3;
5. Documented or suspected liver disease (including laboratory evidence of hepatitis);
6. Recipient of heart transplant;
7. Any patient who previously received murine therapeutic antibodies and exhibited sensitization through the production of Human Anti-murine Antibodies (HAMA);
8. Patient with a life expectancy less than the follow-up period (5 years);
9. Known allergies to aspirin, clopidogrel bisulphate (Plavix®) and ticlopidine (Ticlid®), heparin, or stainless steel;
10. Known side-effects (clinically demonstrated by biological tests, elevated CK and liver assessments) to statins and previous attempts to treat side-effects were unsuccessful;
11. Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study;
12. Currently participating in an investigational drug or another device study that has not completed the primary endpoint, or subject to inclusion in another investigational drug or another device study during follow-up of this study;
13. Patients currently undergoing chemotherapy or immunosuppressant therapy;
14. Patients with known malignancy(ies).

    Angiographic exclusion criteria:
15. Unprotected left main coronary artery disease with ≥ 50% stenosis;
16. Ostial target lesion;
17. Totally occluded target vessel (TIMI flow 0);
18. Target lesion has excessive tortuosity unsuitable for stent delivery and deployment;
19. Target lesion involves bifurcation class D & type G including a side branch ≥ 2.5mm in diameter (either stenosis of both main vessel and major side branch or stenosis of just major side branch) that would require stenting of diseased side branch;
20. Angiographic evidence of thrombus in the target vessel;
21. A significant (> 50%) stenosis proximal or distal to the target lesion;
22. Impaired runoff in the treatment vessel with diffuse distal disease;
23. Ejection fraction ≤ 30%;
24. Pre-treatment with devices other than balloon angioplasty, although direct stenting is allowed;
25. Prior stent within 5mm of target lesion;
26. Intervention of another lesion within 6 months before or within the scheduled angiographic follow-up of the index procedure.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-08; Primary Completion 2008-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is in-stent late loss by Quantitative Coronary Angiography (QCA). | at 6 months

SECONDARY OUTCOMES:
Angiographic success. | during procedure
Procedure success. | during the index hospitalization
Angiographic and/or clinical stent thrombosis. | Up to 5 years
In-stent late loss | at 18 months.
Binary restenosis rate | at 6 and 18 months.
In-segment late loss. | at 6 and 18 months
Volumetric assessment (derived from QCA parameters). | at 6 and 18 months
Circulating endothelial progenitor cell (EPC) count | at screening, index procedure and at 30 days.
Target Vessel Failure (TVF) | at 30 days, 6, 12, 18 months and at 2, 3, 4 and 5 years.
Major adverse cardiac events (MACE) | at 30 days, 6, 12, 18 months and at 2, 3, 4 and 5 years.
Clinically-driven Target Lesion Revascularization (TLR) free rate | at 30 days, 6, 12 and 18 months and at 2, 3, 4 and 5 years.
Protocol related serious adverse events (SAEs) | up to 5 years.
Change in human anti-murine antibody (HAMA) plasma levels | at 1 and 6 months follow-up as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (15):
- Medizinische Universitätsklinik, Graz, Austria
- Belgium (4):
  - OLV Ziekenhuis Aalst, Aalst
  - AZ Middelheim, Antwerp
  - University Hospital Antwerp, Edegem
  - Virga Jesse Ziekenhuis, Hasselt
- Hôpital Henri Mondor, Créteil, France
- Germany (3):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Internistische Klinik Dr. Müller, Munich
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
- United Kingdom (2):
  - Kings College Hospital, London
  - John Radcliflfe Hospital, Oxford

REFERENCES:
- [Derived] den Dekker WK, Houtgraaf JH, Onuma Y, Benit E, de Winter RJ, Wijns W, Grisold M, Verheye S, Silber S, Teiger E, Rowland SM, Ligtenberg E, Hill J, Wiemer M, den Heijer P, Rensing BJ, Channon KM, Serruys PW, Duckers HJ. Final results of the HEALING IIB trial to evaluate a bio-engineered CD34 antibody coated stent (GenousStent) designed to promote vascular healing by capture of circulating endothelial progenitor cells in CAD patients. Atherosclerosis. 2011 Nov;219(1):245-52. doi: 10.1016/j.atherosclerosis.2011.06.032. Epub 2011 Jun 25. PMID 21763653